CLINICAL TRIAL: NCT05838079
Title: Copenhagen Baby Heart Study - Impact
Acronym: CBHS-I
Status: Recruiting | Type: Observational
Sponsor: Henning Bundgaard (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Henning Bundgaard, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-19038069
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous and/or umbilical cord blood sample for DNA extraction and analysis of biomarkers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- New-borns (CBHS-I): New-borns, within the first 30 days of birth.
  Interventions: Other: Clinical examination
- Children (CBH and CBHS-I): Children, 3-13 years of age. The children from the original inclusion in CBH, and those included in CBHS-I.
  Interventions: Other: Clinical examination
- Family members: Children and adults, age 1-99 years of age. Some subprojects will invite the family members of the participating child for family examinations.
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination — Echocardiography Electrocardiography Analysis of umbilical and/or venous blood. Peripheral measurement of oxygen saturation

SUMMARY:
Copenhagen Baby Heart Study - Impact (CBHS-I) is an extension to Copenhagen Baby Heart (CBH) which included over 25.000 new-borns in the Copenhagen area between 2016-2018.

Based on clinical and subclinical deviations in the examinations in CBH, subgroups of participants will be invited to clinical examinations (echocardiography and electrocardiogram) in early childhood. There will also be a new, targeted inclusion based on certain exposures during pregnancy.

The main objectives are to assess the prevalence of congenital and inherited heart disease and, and the development of these during early childhood; examining the association between pre- and postnatal exposure, disease, lifestyle, environmental and genetic factors; continue to establish reference values for echocardiography in Danish neonates and children.

DETAILED DESCRIPTION:
Copenhagen Baby Heart Study - Impact (CBHS-I) is an extension to Copenhagen Baby Heart (CBH) which included over 25.000 new-borns in the Copenhagen area between 2016-2018.

Purpose:

1. To assess the prevalence of congenital and inherited heart disease not detected prenatally, and through follow-up asses the consequence of these, e.g., bicuspid aortic valve and septal defects.
2. To assess the prevalence of structural and functional anomalies detected by echocardiography and electrocardiography shortly after birth and, by follow-up examination, assess the consequence of these in early childhood.
3. To establish reference values for echocardiography and ECG for Danish children.
4. To assess the association between high-risk pregnancies and complications during pregnancy (e.g., twin/multiple pregnancy, assisted human reproduction, preeclampsia, and gestational diabetes) and the risk for congenital heart disease in the offspring and early childhood.
5. To assess the association between maternal chronic diseases (e.g., thyroid disorders or pre-existing diabetes) and the risk for congenital heart disease in the offspring and early childhood.
6. To assess the life-long development of cardiovascular disease as well as other conditions and to study associations between both pre- and postnatal exposure and disease, including lifestyle, environmental and genetic factors.

Methods The birth cohort of CBH constitute over 25.000 new-borns. At birth an umbilical cord blood sample was taken and immediately analysed for routine biochemical markers, and samples were also stored for possibility of future analyses and DNA sequencing.

All clinical examinations (echocardiography, electrocardiography, and measurement of oxygen saturation) took place within the first 2nd month of life, the vast majority within the 1st month, median age at examination was 11 days (interquartile range 7-15). In addition to this CBH has built a unique and extended database which include information about the maternal and paternal health, the pregnancy and birth.

As part of CBHS-I subgroups of the CBH cohort (e.g., children born to mothers with diabetes or preeclampsia, or children with abnormal findings at baseline examinations in CBH) will be invited for follow-up examinations (echocardiography and electrocardiography). There will also be a new inclusion of new-borns from the same geographical area and Hospitals as in CBH in order to expand some of the sub cohorts, e.g., children born to mothers with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participant in CBH or
* Family member of a participant in CBH or
* Born to mothers with pre-existing or gestational diabetes at either Rigshospitalet, Hvidovre Hospital, or Herlev Hospital during the period July 2020 through December 2023.

Exclusion Criteria:

* Faliure of providing concent (parents)

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants from CBH and in some cases their family members. New-borns of mothers with pre-existing or gestational diabetes, included during CBHS-I.
Sampling Method: Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of congenital heart disease | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bundgaard, MD, DMSc, Principal Investigator — Department of Cardiology, The Heart Center, Rigshospitalet, Copenhagen University Hospital, Denmark; Kasper Iversen, MD, DMSc, Principal Investigator — Department of Cardiology, Herlev Hospital, Denmark.
Locations (3):
- Denmark (3):
  - Rigshospitalet Copenhagen University Hospital., Copenhagen Ø
  - Herlev and Gentofte Hospital, Herlev
  - Hvidovre Hospital, Hvidovre